CLINICAL TRIAL: NCT06548061
Title: Single Center Observational Study Using Spinal Laser Interstitial Thermal Therapy (sLITT) in the Treatment of Spine Metastases and Tumors
Brief Title: D20054;LITT for Spine Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Linton T. Evans, Director, Neuro-oncology, Principle Investigator, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001761
Record Dates: First submitted 2023-03-09; First posted 2024-08-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Spinal Metastases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spinal Laser Interstitial Thermal Therapy (sLITT) (Experimental): Patients will undergo surgery utilizing the Visualase Thermal Therapy System (Medtronic) device.
  Interventions: Device: ClearPoint Prism

INTERVENTIONS:
Device: ClearPoint Prism — Spine laser interstitial therapy used instead of open decompression followed by spine stereotactic radiosurgery (SSRS).

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety of spinal laser interstitial therapy in the treatment of metastatic spinal tumors. The investigators hypothesize that rates of local tumor control are comparable between conventional open surgical techniques and spinal laser interstitial therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histology confirmed spinal tumor involving the T2-T12 spine segments.
2. Indication for spine stereotactic radiosurgery or palliative intervention.
3. Normal neurologic exam at the time of presentation (Frankel grade E).

Exclusion Criteria:

1. Contraindication to MRI
2. ANY neurologic deficit
3. Tumor spanning more than 3 consecutive vertebral segments
4. Contraindication to general anesthesia
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Local tumor control | Local control rate at 12 months
  Any increase in the epidural spinal cord compression score (ESCC grade 1 (no compression) to 3 (spinal cord compression) compared to the initial post-procedure MRI will be considered local radiographic failure or evidence of tumor recurrence.

SECONDARY OUTCOMES:
Evaluate neurologic function before and after sLITT. | 3, 6, 9, and 12 months post-operatively
  Using Frankel score. Frankel scores (scale form A to E where A= complete loss of motor and sensory function, B= complete motor paralysis but some sensory function, C= some motor function but not usable, D= weakened but usable motor function, E= neurologically intact)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Health, Lebanon, New Hampshire, United States